CLINICAL TRIAL: NCT01657253
Title: A Randomized, Double-blind, Phase III Clinical Trial to Evaluate the Efficacy and Safety of PRO-148 Versus Systane®, in Patients With Mild to Moderate Dry Eye
Brief Title: Efficacy and Safety of PRO-148 Versus Systane®, in Patients With Mild to Moderate Dry Eye
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SOPH148-0512/III
Record Dates: First submitted 2012-07-19; First posted 2012-08-06 (Estimated); Results first posted 2017-12-15 (Actual); Last update posted 2017-12-15 (Actual); Status verified 2017-05

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — xanthan gum; Chondroitin; Propylene Glycol; hydroxypropyl guar

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PRO-148 (Experimental): PRO-148 containing: xanthan gum and sulphate chondroitin, ophthalmic solution
  doses: 1 drop in each eye, quarter in day
  Interventions: Drug: PRO-148
- Systane® (Active Comparator): Systane containing: polyethylene glycol 400 0.4%, propylene glycol 0.3% and hydroxypropyl guar
  doses: 1 drop in each eye, quarter in day
  Interventions: Drug: Systane

INTERVENTIONS:
Drug: PRO-148 — Instill 1 drop in each eye four times a day, for 60 days
  Other Names: PRO-148 (xanthan gum and sulphate chondroitin)
  Arms: PRO-148
Drug: Systane — Instill 1 drop in each eye four times a day, for 60 days
  Other Names: polyethyleneglycol 400, propyleneglycol, hydroxypropyl guar
  Arms: Systane®

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of the ophthalmic solution PRO-148 in the ocular surface of patients with mild to moderate dry eye compared with ophthalmic solution Systane®

DETAILED DESCRIPTION:
Dry eye is a multifactorial disease of the tears and ocular surface that results in symptoms of discomfort, visual disturbance, and tear film instability with potential damage to the ocular surface. Current treatment is heavily weighted toward supplementation, stimulation, or preservation of aqueous tears. Artificial tears are one of the primary treatments for dry eye; it is mainly palliative and focuses on reducing the symptoms of discomfort to improve quality of life for a patient.

A phase III randomized double-blind clinical trial will be conducted to evaluate efficacy and safety of the ophthalmic solution PRO-148 in the ocular surface of patients with mild to moderate dry eye compared with ophthalmic solution Systane®. Patients will be randomized to receive one of the treatments for 60 days. Efficacy and safety measures will be performed at baseline and at 60 days after treatment

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate dry eye patients based on the Report of International Dry Eye Workshop (DEWS)
* OSDI score between 12 and 45
* Provided informed consent

Exclusion Criteria:

* Patients with one blind eye
* Visual acuity of 20/100 or worst in any eye
* Patients with any active ocular disease that would interfere with study interpretation
* Patients in treatment with any medication that could interfere with the study, contraindication of any medication used in the protocol
* Patients with history of hypersensitivity or contraindication for any drug used in the study
* Contact lens users
* Pregnant patients, at risk of pregnancy or breastfeeding
* Patients without birth control treatment
* Patients who had participated in any clinical trial in the last 90 days
* Legal or mentally disabled patients who could not give informed consent
* Patients who do not provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2013-11; Primary Completion 2015-02 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leopoldo M Baiza-Durán, MD, Study Director — Laboratorios Sophia S.A de C.V.
Locations (1):
- Consultorio privado, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No
The personal data of the study subjects were treated with Confidentiality policy.

REFERENCES:
- [Derived] Perez-Balbuena AL, Ochoa-Tabares JC, Belalcazar-Rey S, Urzua-Salinas C, Saucedo-Rodriguez LR, Velasco-Ramos R, Suarez-Sanchez RG, Rodriguez-Carrizalez AD, Oregon-Miranda AA. Efficacy of a fixed combination of 0.09 % xanthan gum/0.1 % chondroitin sulfate preservative free vs polyethylene glycol/propylene glycol in subjects with dry eye disease: a multicenter randomized controlled trial. BMC Ophthalmol. 2016 Sep 20;16(1):164. doi: 10.1186/s12886-016-0343-9. PMID 27645318

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period started since february 2014 to january 2015. sites of research: Private Medical Office, Ophthalmology Hospitals (nationals and internationals)
  Patients with:
  * mild to moderate Dry eye
  * age > 18 year old
  * OSDI between 12 and 45
  * TBUT ≤ 10 seconds
  * Schirmer test ≤ 10mm
Pre-assignment Details: 183 patients were enrolled at baseline, however, only 148 ended the period of intervention and 35 were excluded or deleted by different reasons.
Groups:
- PRO-148: PRO-148 containing: xanthan gum and sulphate chondroitin, ophthalmic solution
  doses: 1 drop in each eye, quarter in day
  PRO-148: Instill 1 drop in each eye four times a day, for 60 days
- Systane®: Systane containing: polyethylene glycol 400 0.4%, propylene glycol 0.3% and hydroxypropyl guar
  doses: 1 drop in each eye, quarter in day
  Systane: Instill 1 drop in each eye four times a day, for 60 days
Period: Overall Study
Arm/Group | PRO-148 | Systane®
Started | 93 | 90
Completed | 76 | 72
Not Completed | 17 | 18
Not completed — Lost to Follow-up | 6 | 5
Not completed — Withdrawal by Subject | 11 | 12
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: The comparative between baseline and final characteristics, in this section, is considering patients with completely evaluation
Groups:
- Total: Total of all reporting groups
Arm/Group | PRO-148 | Systane® | Total
Number analyzed (Participants) | 93 | 90 | 183
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.3 (16.0) | 45.3 (13.8) | 46.8 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 65 | 132
  Male | 26 | 25 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 93 | 90 | 183
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 59 | 63 | 122
  Chile | 17 | 15 | 32
  Colombia | 17 | 12 | 29

OUTCOME MEASURES:

1. Primary Outcome: Ocular Surface Disease Index (OSDI©) Questionnaire
Description: Ocular Surface Disease Index (OSDI©) questionnaire , consists of 12 questions divided in 3 groups, Each question has a value that can go from 0 to 4 points according to the severity of the case: 0.None of the time, 1. Some of the time, 2.Half of the time, 3.most of the time and 4 all of the time. The points of all the questions will be used in the following formula for converted to a score of 0-100 : (sum of scores) x 25 / (# of questions answered), where 0 represents normality or non-symptomatology and 100 the most severe case. Will be used to measure the symptoms of dry eye disease by obtaining baseline data and comparing them against the last visit.
Time Frame: Day 60
Measure: Mean (Standard Deviation); unit: points
Units Other Than Participants: eyes
Arm/Group | PRO-148 | Systane®
Number analyzed (Participants) | 76 | 72
Number analyzed (eyes) | 152 | 144
points
  baseline values | 19.3 (7.4) | 19.3 (7.5)
  final values | 7.3 (5.9) | 7.9 (8.2)

2. Secondary Outcome: Schirmer Test
Description: Change from Baseline in Schirmer test after 60 days of treatment
  Schirmer test
  It is the technique most used to measure aqueous and at the same time the simplest tear secretion. It is carried out as follows: Without applying anesthesia, the patient is placed somewhere without much illumination, without applying anesthesia, a strip of filter paper of approximately 30 mm is placed, of which, 5 mm must go in the joint Of the middle and outer third of the lower eyelid. The patient is instructed to look forward and to blink normally. After 5 minutes the strips are removed and the wetting is recorded in millimeters. A test less than or equal to 6 mm is diagnostic of aqueous deficiency.The mean of the revisions by group will be compared at the baseline and final visit.
Time Frame: Day 60
Measure: Mean (Standard Deviation); unit: mm/min
Units Other Than Participants: eyes
Arm/Group | PRO-148 | Systane®
Number analyzed (Participants) | 76 | 72
Number analyzed (eyes) | 152 | 144
mm/min
  baseline values | 6.4 (2.2) | 6.5 (2.5)
  final values | 11.0 (6.6) | 10.5 (5.6)

3. Secondary Outcome: Tear Film Break up Time
Description: Change from Baseline in Tear film break up time after 60 days of treatment Tear film breakup time is the elapsed time from blinking to the first occurrence of a dry area in the cornea, visualized with the help of fluorescein staining. Measurement of tear film breakup time will be performed as follows: Fluorescein is instilled in the eye, the patient is asked to blink three times to distribute the dye and then set the eye to the front and do not blink while the examiner observes the cornea with cobalt blue light, looking for an area of tear film rupture, which is manifested by the appearance of a black island within the fluorescein green film. Normally film breakup time is 10 seconds or more and the minimum register may be 1 second, Under 10 seconds is considered abnormal.
Time Frame: Day 60
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: eyes
Arm/Group | PRO-148 | Systane®
Number analyzed (Participants) | 76 | 72
Number analyzed (eyes) | 152 | 144
seconds
  baseline values | 5.5 (2.1) | 5.2 (2.0)
  final values | 7.4 (2.9) | 7.4 (2.7)

ADVERSE EVENTS:
Time Frame: The evaluation of serious and no serious adverse events was done during 15 months
Description: in each clinical visit, the ophthalmologist completed the case report and the adverse events format
Arm/Group | PRO-148 | Systane®
Serious Adverse Events (participants affected / at risk) | 0/93 | 1/90
Other Adverse Events (participants affected / at risk) | 14/93 | 5/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRO-148 (N=93) | Systane® (N=90)
heart attack (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRO-148 (N=93) | Systane® (N=90)
Conjunctivitis (Eye disorders) | 5 (5) | 0 (0) — During the study 5 patients reported conjunctivitis: 2 patients with allergic conjunctivitis 1. patient with bacterium conjunctivitis 2. patients with acute nonspecific conjunctivitis
ocular burning sensation (Eye disorders) | 3 (3) | 0 (0) — During the study, 3 patients reported ocular burning sensation
Pruritus (Eye disorders) | 2 (2) | 0 (0) — In the systematic evaluation, 2 patients reported pruritus
Red eye (Eye disorders) | 1 (1) | 0 (0) — In the systematic evaluation, 1 patient presented red eye
rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) — During the evaluation, 4 patients had rhinitis.
Back spasm (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — 1 patient refered back spasm during his participation in the present study
Dental extraction (Surgical and medical procedures) | 1 (1) | 0 (0) — 1 patient had infection in one piece dental during his participation in this study
Lower back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — 1 patient had lower back pain during its participation in the present study
Change in the visual acuity (Eye disorders) | 0 (0) | 1 (1) — 1 patient in the PRO-148 group reported change in the visual acuity. When the clinical ophthalmologist reviewed to the patient, the visual acuity was good.

LIMITATIONS AND CAVEATS:
The study was performed according to the clinical protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All the information is confidential and exclusive property of the sponsor. Information can be revealed only to my staff and regulatory agencies or ethics committee.

All the information from this protocol is confidential and exclusive property of the sponsor, it can not be revealed without written consent from the sponsor.